CLINICAL TRIAL: NCT00087841
Title: Midcareer Development of Nonpharmacologic Analgesia
Brief Title: Self-Hypnotic Relaxation Therapy During Invasive Procedures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K24AT001074-01 (NIH)
Record Dates: First submitted 2004-07-14; First posted 2004-07-16 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Uterine Neoplasms; Leiomyoma
Keywords: Hypnosis; Analgesia; Embolization, Therapeutic; Chemoembolization, Therapeutic
MeSH Terms: conditions — Uterine Neoplasms; Leiomyoma; Agnosia

INTERVENTIONS:
Behavioral: Self-hypnotic relaxation

SUMMARY:
The purpose of this study is to determine the effectiveness of self-hypnotic relaxation on mental and physical distress during and after tumor treatment procedures.

DETAILED DESCRIPTION:
Pain relievers and sedatives may have limited effectiveness and serious side effects when given to alleviate distress during minimally invasive surgical procedures. Unabated distress may interfere with the ongoing procedure and may negatively impact future interventions.

Studies have shown that nonpharmacologic analgesia in the form of self-hypnotic relaxation during invasive medical procedures significantly reduces patients' pain, anxiety, drug use, and number of complications. The long-term goal of this study is to determine whether self-hypnotic relaxation therapy can be a safe and practical method for reducing cognitive and physiologic distress associated with invasive procedures.

Participants in this study will be randomly assigned to one of three groups: a standard care group, an empathic control group, and a self-hypnotic relaxation group. The emphatic control group will meet with a clinician who will offer encouragement and support. The group assigned to self-hypnotic relaxation will read a standardized script prior to procedure. Self-report questionnaires will be used to assess pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Referred for transcatheter embolization for benign uterine fibroid tumor or radiofrequency ablation or chemoembolization for malignant tumors
* Able to hear and understand English

Exclusion Criteria:

* Impaired mental function
* Psychosis
* Severe chronic obstructive pulmonary disease
* Intolerance of midazolam or fentanyl
* Weigh less than 121 lbs
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390
Dates: Start 2002-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Lang, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States